CLINICAL TRIAL: NCT07141823
Title: Oxidative DNA Damage Enhancement by Vitamin C Among Narghile Smokers and Non-smokers
Acronym: DNA Damage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nora Tariq Mohammed (Other)
Responsible Party: Sponsor-Investigator, Nora Tariq Mohammed, MSc Student in Biochemistry, University of Duhok
Organization: University of Duhok (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: UoD-ODNS-2025-01
Record Dates: First submitted 2025-07-16; First posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-07

CONDITIONS: Narghile
Keywords: DNA damage, Oxidative stress ,MDA; vitamin C
MeSH Terms: conditions — Water Pipe Smoking | interventions — Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Narghile nonsmokers vitamin C taking (Experimental): this group of participant take vitamin C for one month, and they are healthy volunteers
  Interventions: Dietary Supplement: Vitamin C (Ascorbic Acid) regularly has been taken
- Narghile smokers (Experimental): this group take vitamin c supplent for one month period and are healthy.
  Interventions: Dietary Supplement: Vitamin C (Ascorbic Acid) regularly has been taken

INTERVENTIONS:
Dietary Supplement: Vitamin C (Ascorbic Acid) regularly has been taken

SUMMARY:
This study aims to evaluate oxidative DNA damage among hookah smokers compared to non-smokers by measuring biomarkers of oxidative stress in blood samples. The objective is to determine the impact of hookah smoking on DNA integrity and overall oxidative status in adults.

DETAILED DESCRIPTION:
Hookah smoking has become increasingly popular in many regions, yet its potential impact on oxidative stress and DNA integrity is not fully understood. This study aims to investigate the level of oxidative DNA damage among hookah smokers compared to non-smokers by analyzing biomarkers in blood samples. A case-control observational design will be used, involving two groups of adult participants: regular hookah smokers and age-matched non-smokers. Blood samples will be collected from all participants and analyzed for markers of oxidative stress, including 8-hydroxy-2'-deoxyguanosine (8-OHdG) and malondialdehyde (MDA), using validated biochemical methods. The findings are expected to provide insights into the biological consequences of hookah smoking and support the development of public health interventions.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-30 years

Current narghile (hookah) smokers for at least 1 year

Willing to provide informed consent

Exclusion Criteria:

* Healthy participant

Ages: 18 Months to 30 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 96 (Actual)
Dates: Start 2024-10-15 (Actual); Primary Completion 2024-12-10 (Actual); Study Completion 2025-03-10 (Actual)

PRIMARY OUTCOMES:
Oxidative DNA damage | Baseline and after 1 month
  Measurement of plasma MDA concentration using the thiobarbituric acid reactive substances (TBARS) method to assess oxidative stress in participants before and after 1-month Vitamin C supplementation and measuring oxidative stress marker and TAOC

CONTACTS AND LOCATIONS:
Locations (1):
- University of Duhok, Duhok, semel, Iraq